CLINICAL TRIAL: NCT04748224
Title: Evaluation of the Analgesic Efficacy of Dexmedetomidine as an Adjuvant to Local Anesthesia in Quadratus Lumborum Block After Cesarean Delivery: A Randomized Controlled Trial.
Brief Title: Dexmedetomidine as an Adjuvant to Local Anesthesia in Quadratus Lumborum Block After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed elaraby, assistant lecturer of anesthesia,icuand pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MD-75-2020
Record Dates: First submitted 2021-01-15; First posted 2021-02-10 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, investigators, care providers and outcome assessors will be blinded to the study group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (bupivacaine only) (Active Comparator): Group A will be injected with 20 ml of 0. 25% bupivacaine in each side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- group B (bupivacaine plus dexmedetomidine) (Active Comparator): Group B will be injected with 20 ml of 0. 25% bupivacaine in each side added to it dexmedetomidine 0.5 μg/kg; (Precedex 100 μg/ml (Hospira, inc, lake forest, USA).
  Interventions: Drug: bupivacaine plus dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — a local anesthetic drug
  Other Names: marcaine
  Arms: group A (bupivacaine only)
Drug: bupivacaine plus dexmedetomidine — bupivacaine is a local anesthetic drug plus dexmedetomidine is a new generation highly selective α2-adrenergic receptor (α2-AR) agonist that is associated with sedative and analgesic sparing effects
  Other Names: Marcaine plus precedex
  Arms: group B (bupivacaine plus dexmedetomidine)

SUMMARY:
Postoperative pain is considered one of the major problems after abdominal operations, so proper pain control is one of the main issues in clinical practice. Cesarean section (CS.) is one of the most common abdominal surgeries and the use of CS. worldwide has increased to unprecedented levels. Effective postoperative analgesia enhances early recovery of the delivered mother, early ambulation, breast feeding and decreases the risk of postoperative thromboembolism. Therefore, Opioids are prescribed routinely for postoperative pain control, but they have many adverse effects such as nausea, vomiting, constipation, excessive sedation, dizziness, respiratory depression, and addiction, so it is important to practice alternative opioid sparing analgesic approaches. Recently, QL block is considered one of the perioperative pain management techniques used in patients undergoing various pelvi-abdominal surgeries. Quadratus Lumborum block inhibits both pain components (somatic and visceral) as a result of local anesthetic spread to the paravertebral spaceA study has been published comparing the analgesic efficacy between QLB and TAP block after cesarean section and proved that QL block II is more effective than TAP Block regarding pain relief and duration of action after CS. Also, Many studies have been published and prove that Combination of adjuvants like (fentanyl, clonidine and MgSo4,etc.) to local anesthetics agents helps in prolonging the analgesic effect and decrease 24hours opiate consumption.one of these adjuvants which used extensively in the regional techniques is dexmedetomidine, which is a selective alpha-2 adrenergic agonist. The optimal dosage of dexmedetomidine to be added to local anesthetics still remains unclear, but in other studies the dose of 0.5 μg/kg is widely used with no postoperative complications.

in this double blinded randomized controlled trial, the investigators compare the analgesic efficacy of adding dexmedetomidine to local anesthetic in quadratus lumborum block and their role in reduction postoperative opioid consumption after cesarean section

DETAILED DESCRIPTION:
Using a computer-generated randomization schedule, fifty patients will be randomly assigned into two equal groups: group A (bupivacaine only; n=25) and group B (bupivacaine plus dexmedetomidine; n=25).

All participants, investigators, care providers and outcome assessors will be blinded to the study group allocation.

The day Prior to surgery, all patients will have pre anesthesia check-up with routine and subjective investigations and explained about the Numerical Rating Scale (NRS) ranging from 0-10 (0 indicating no pain and 10 for severe intractable pain) The patients will be pre medicated by 40mg oral pantoprazole at night and in the morning of the surgery.

On arrival to the operating room, patients will be monitored by peripheral pulse oximetry, five-lead electrocardiogram and non-invasive blood pressure monitor. Two 18-gauge intravenous cannulae will be inserted in the nondominant arm and 1500 ml crystalloid will be infused as acoload plus ephedrine infusion 4mg/min. to prevent post spinal hypotension.

Random allocation of patients into one of two groups using concealed closed envelope method, the patients' envelope which contain the number of group will be opened and recorded in the data collection sheet as a number of group because the data collector will be blinded to the intervention on the patient, only the anesthetist knows each number is referring to which intervention.

Spinal anesthesia will be performed with the patient in the sitting position at the level of L2 to 3 or L3 to 4 intervertebral spaces using a 25-gauge Quincke Bevel type needle (Spinocan®, Braun Melsungen AG,Germany) with 10 mg of hyperbaric bupivacaine(AstraZeneca Pharmaceuticals, UK) and 25μ g of fentanyl. Patients will be placed in the supine position with left uterine displacement and a face-mask will be applied to deliver oxygen at rate of 6 L/minute.

Five minutes after spinal injection, Spinal anesthesia level will be assessed by loss of cold (ice cube) and touch (blunt pin) discrimination and will be considered successful if a bilateral sensory blockade to T4-T6 is established. Anesthesia and surgical management will be performed in the usual manner.

At the end of surgery, all patients will receive 1 gm of intravenous paracetamol. After the abdomen will be cleaned with surgical solution, covering the wound and while the patient is still fully monitored, the patient will be placed in the lateral decubitus position and the QLB will be performed.

A convex (5-8 MHz) ultrasound probe (Shenzhen Mindray BIO-Medical Electronics, Model: DP-20, China) with a protective sheath will be used after imaging depth and gain is adjusted. The procedure will be done under complete aseptic condition (facemask, gown, and gloves) after cleaning of the abdominal skin with antiseptic solution.

The probe will be placed in the mid axillary line cranially to the iliac crest to identify the three muscles of the anterior abdominal wall (transversus abdominis, internal oblique, and external oblique). Then, scan dorsally keeping the transverse orientation until observing that the transversus abdominus muscle became aponeurotic, and this aponeurosis will be followed until the QL muscle is clearly visualized with its attachment to the lateral edge of the transverse process of the L2 vertebral body and visualize the thoracolumbar fascia at the lateral edge of the QL muscle , followed by recognition of Shamrock pattern by viewing psoas major muscle (PM) anteriorly, the erector spinae muscle (ESM) posteriorly and the QL muscle adherent to the apex of the transverse process (trifoliate).

Stimuplex® A 21G 100-mm needle (B. BRAUN, Melsungen AG, Germany) will be inserted in plane under real time US guidance from anterolateral to posteromedial direction via the abdominal wall. Two milliliters of 0.9% saline will be injected to visualize the solution spread (hydro dissection) to determine the optimal point of injection over the lumbar interfacial triangle.

Group A will be injected with 20 ml of 0. 25% bupivacaine in each side. (14) Group B will be injected with 20 ml of 0. 25% bupivacaine in each side added to it dexmedetomidine 0.5 μg/kg; (Precedex 100 μg/ml (Hospira, inc, lake forest, USA).

Patients will be transferred to the post anesthesia care unit (PACU) and discharged from PACU when fully conscious, hemodynamically stable and pain free.

All patients will receive IV paracetamol 1gm every 8 hours. As a rescue analgesic, IV morphine (0.05 mg/kg) will be given when Numerical Rating Scale (NRS) > 3, maximum dose of morphine will be given 30 mg per day.

the following data will be recorded:

* Total morphine consumption at predetermined time intervals (4, 8, 12, and 24) hrs. after surgery
* Numerical Rating Scale (NRS) ranging from 0-10 (0 indicating no pain and 10 for severe intractable pain) will be recorded and compared at 4,8,12, and 24h after surgery.
* Incidence of post-operative complications as nausea, vomiting or abdominal distension will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for cesarean section under spinal anesthesia.
2. Normal uncomplicated pregnancies (ASA II).
3. BMI 18.5 to 34.9 kg/m2

Exclusion Criteria:

1. Patient refusal.
2. ASA III - IV patients.
3. Coagulation disorders.
4. Skin lesions or infection at site of proposed needle.
5. Known allergy to any of study drugs.
6. inability to comprehend or use the verbal rating pain scoring system
7. Difficulty in Ultrasonographic identification.
8. Opioid abuse.
9. BMI > 35 Kg/m2.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
total amount of morphine consumption | up to 24 hours
  Measure the total amount of morphine consumption at predetermined time intervals (4, 8, 12, and 24) hrs. after surgery

SECONDARY OUTCOMES:
Numerical Rating Scale | up to 24 hours
  Numerical Rating Scale at rest (static), and on movement (dynamic) at 4, 8, 12, and 24 hours postoperatively.
  it requires the patient to rate their pain on a defined scale from 0 to 10 where 0 is no pain and 10 is the worst pain imaginable

OTHER OUTCOMES:
ambulation postoperatively | up to 24 hours
  Time to first Ambulation postoperatively
quadratus lumborum block complications | up to 24 hours
  Quadratus lumborum Block related complications e.g. bowel injury, hematoma formation, nerve injury and intravascular injection.
sedation score | up to 24 hours
  Sedation scores (Ramsay scale), itching (0, none; 1, mild; 2, moderate; and 3, severe), nausea (0, none; 1, mild;2, moderate; and 3, severe or vomiting), and other complications postoperatively
Postoperative side effects related to dexmedetomidine | up to 24 hours
  Postoperative side effects related to dexmedetomidine e.g. bradycardia and hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrine M. El-Refai, professor, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Medicine Cairo University, Cairo
  - Faculty of Medicine, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Snell P, Hicks C. An exploratory study in the UK of the effectiveness of three different pain management regimens for post-cesarean section women. Midwifery. 2006; 22(3):249-61. 2. Betrán A, Ye J, Moller A, et al. The Increasing Trend in Cesarean Section Rates: Global, Regional and National Estimates: 2016;11(2) 3. Gadsden J, Hart S, Santos A. Post-cesarean delivery analgesia. Anesth Analg 2005; 101(5 Suppl): S62-S69. 4. Karlström A, Engström-Olofsson R, Norbergh K, et al. Postoperative pain after cesarean birth affects breastfeeding and infant care. J Obstet Gynecol Neonatal Nurs 2007; 36: 430-40. 5. Stephan B, Parsa F. Avoiding Opioids and Their Harmful Side Effects in the Postoperative Patient: Exogenous Opioids, Endogenous Endorphins, Wellness, Mood, and Their Relation to Postoperative Pain. Hawai'i journal of medicine & public health: a journal of Asia Pacific Medicine & Public Health. 2016 Mar; 75(3):63-7. 6.Mieszkowski M, Zawadzka E, Tuyakov B, et al. Evaluation of the effectiveness of the Quadratus Lumborum Block type I using ropivacaine in postoperative analgesia after a cesarean section - a controlled clinical study. Ginekologia Polska 2018; 89: 89-96. 7. Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after cesarean section: a randomized controlled trial. Eur J Anesthesiol. 2015; 32: 812-8. 8. Blanco R, Ansari T, Riad W, et al. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016; 41: 757-62. 9. Singh R, Kumar N, Jain A, et al. Addition of clonidine to bupivacaine in transversus abdominis plane block prolongs postoperative analgesia after cesarean section. J Anesthesiol ClinPharmacol 2016; 32:501-4. 10. Sarvesh B, Shivaramu B, Sharma K, et al. Addition of Dexmedetomidine to Ropivacaine in Subcostal Transversus Abdominis Plane Block Potentiates Postoperative Analgesia among Laparoscopic Cholecystectomy Patients: A Prospective Randomized Controlled Trial. Anesth Essays Res. 2018; 12(4):809-813. 11.Kirksey M, Haskins S, Cheng J, et al. Local Anesthetic Peripheral Nerve Block Adjuvants for Prolongation of Analgesia: A Systematic Qualitative Review. PLoS One. 2015; 10(9). 12. Varshney A, Prabhu M, Periyadka B, et al. Transversus abdominis plane (TAP) block with levobupivacaine versus levobupivacaine with dexmedetomidine for postoperative analgesia following cesarean delivery. J Anesthesiol Clin Pharmacol. 2019; 35(2):161-164. 13- Qianchuang S, Shuyan L, Huiying u, et.al. Dexmedetomidine as an Adjuvant to Local Anesthetics in Transversus Abdominis Plane Block. A Systematic Review and Meta-analysis Clin J Pain. 2019 Apr; 35(4): 375-384. 14. Carline L, McLeod G, Lamb C. A cadaver study comparing spread of dye and nerve involvement after three different quadratus lumborum blocks. Br J Anesth. 2016; 117(3):387-394. 15. Kılıç E, Bulut E. Quadratus Lumborum Block III for Postoperative Pain AfterPercutaneous Nephrolithotomy. Turk J Anesthesiol Reanim. 2018; 46(4):272-275.